CLINICAL TRIAL: NCT06673368
Title: A Phase 2 Randomized Double-Blind, Parallel, Adaptive-Design, Clinical Trial to Evaluate the Safety and Efficacy of NRCT-101SR With NRCT-202XR Compared to NRCT-202XR Alone in Subjects With Attention-Deficit/Hyperactivity Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Neurocentria, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NC-022A
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-03

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: A multi-center, randomized, double-blind, parallel, adaptive-design clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Active Comparator): NRCT-101SR and low dose NRCT-202XR
  Interventions: Drug: NRCT-101SR, NRCT-202XR
- Arm 2 (Active Comparator): NRCT-101SR placebo and high dose NRCT-202XR
  Interventions: Drug: NRCT-101SR, NRCT-202XR
- Arm 3 (Active Comparator): NRCT-101SR placebo and low dose NRCT-202XR
  Interventions: Drug: NRCT-101SR, NRCT-202XR

INTERVENTIONS:
Drug: NRCT-101SR, NRCT-202XR — NRCT-101SR in combination with NRCT-202XR or NRCT-202XR alone

SUMMARY:
A combination therapy of NRCT-101 with NRCT-202 is being developed for patients with ADHD.

DETAILED DESCRIPTION:
A multi-center, randomized, double-blind, parallel, adaptive-design clinical trial to evaluate the safety and efficacy of co-administration of NRCT-101SR and low dose NRCT- 202XR compared to low or high dose of NRCT-202XR and placebo NRCT-101SR over a 6-week period in approximately 60 pediatric subjects (13-17 years of age) with ADHD.

Subjects' enrollment will be conducted in two stages.

In stage 1, subjects are planned to be randomized to one of the following two arms (1:1 ratio):

Arm 1: NRCT-101SR and low dose NRCT-202XR Arm 2: NRCT-101SR placebo and high dose NRCT-202XR

In stage 2, a third study arm will be added (Arm 3 - NRCT-101SR placebo and low dose NRCT-202XR.

The study population will include male and female subjects (sex assigned at birth) of all races/ethnicities with ADHD.

ELIGIBILITY:
1. Male or female, 13-17 years of age at screening.
2. Has a prior primary diagnosis of ADHD according to the DSM-5 classification evident by a medical record and confirmed with MINI using DSM-5 probes.
3. Is taking ADHD medication 4-7 days/week, for at least 4 weeks at Screening and at least 6 weeks at Baseline.
4. Has side effects identified using SDSE-RS at Screening and Baseline.
5. CGI-S ≥ X (blinded) at Screening and Baseline.
6. Must be fluent in English and communicate effectively with others.
7. Both subject and parent/guardian willing and able to give informed assent/consent.
8. Parent/guardian willing to serve as informant.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
CGI-S | 6 weeks
SDSE-RS | 6 weeks

SECONDARY OUTCOMES:
CBRS-P | 6 weeks
  and academic problems in children between the ages of 6 and 18 years and are reported by parents.
DPREMB-R | 6 weeks
ADHD-RS-5 | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Guy Bar-Klein, PhD, Study Director — Neurocentria, Inc.
Locations (5):
- United States (5):
  - Accel Research Site-Maitland Clinical Research Unit, Maitland, Florida
  - iResearch Atlanta, Decatur, Georgia
  - CenExel iRS - iResearch Savannah, Savannah, Georgia
  - Boston Clinical Trials LLC, Boston, Massachusetts
  - Center For Psychiatry and Behavioral Medicine, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No